CLINICAL TRIAL: NCT06040073
Title: Natural History of Coronary Atherosclerosis Based on Multimodal Imaging and Physiological Fusion Techniques (NASCENT)
Brief Title: Natural History of Coronary Atherosclerosis
Acronym: NASCENT
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Lei Song, MD, Director of the Coronary Heart Disease Ward, First Section, China National Center for Cardiovascular Diseases
Other Study IDs: 2023-GSP-GG-3
Record Dates: First submitted 2023-09-03; First posted 2023-09-15 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease Progression; Radial Wall Strain; Atherosclerotic Lesion; Optical Coherence Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study sought to explore the predictive value of radial wall strain (RWS, derived solely from angiograms) for coronary artery lesion progression compared with lesion vulnerability assessed by optical coherence tomography (OCT). The lesion progression at 1 year was defined as an increase of ≥20% in diameter stenosis based on quantitative coronary angiography (QCA) evaluation.

DETAILED DESCRIPTION:
The recently developed angiography-derived maximum RWS (RWSmax) was computed as the maximum deformation of lumen diameter throughout the cardiac cycle, expressed as a percentage of the largest lumen diameter. This approach offers a quantitative assessment of the biomechanical attributes of coronary lesions. Consequently, it allows for the identification of lesion vulnerability, potentially compensating for the limitations of intravascular imaging in assessing lesion stability and optimizing strategies for identifying high-risk vulnerable plaques in patients.

In the present multicenter, prospective cohort of individuals with acute myocardial infarction, we assessed the predictive significance of identifying vulnerable lesions using an RWSmax threshold of ≥13%. The investigation aimed to determine the capacity of these identified lesions to predict the progression of the disease at 1 year. Furthermore, the study validated that predictive capacity of RWSmax was on par with, and not inferior to, lesion vulnerability assessed by OCT in tracking lesion progression.

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion Criteria:

  1. Age ≥18 years
  2. Acute myocardial infarction ≤ 45 days
  3. Planned coronary angiography examination or potential interventional treatment
* Angiographic Inclusion Criteria:

  1. The presence of at least 1 non-flow-restricting lesion (visually estimated diameter stenosis: 30%-80%; QFR > 0.80) in any non-infarct related artery with RVD ≥2.5 mm by visual assessment

Exclusion Criteria:

* General exclusion Criteria:

  1. Cardiogenic shock
  2. Pregnant or woman of child-bearing potential
  3. Life expectancy less than 1 year for non-cardiac causes
  4. Unable to tolerate contrast agents or anticoagulant/antiplatelet therapy
  5. Prior CABG or planned CABG
* Angiographic exclusion Criteria:

  1. Poor angiographic image quality precluding vessel contour detection or with suboptimal contrast opacification, branch ostium cannot be shown clearly, severe overlap in the stenosed segment or severe tortuosity of any interrogated vessel deemed not amenable to QFR or RWS measurement
  2. An interrogated lesion require surgical bypass grafting
  3. Unable to judge culprit lesion or infarct-related artery according to current evidence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult study participants with acute myocardial infarction complicated by multi-vessel coronary artery diseases within 45 days.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-07-07 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Lesion progression assessed by QCA | 1 year
  Defined as an increase of ≥20% in diameter stenosis based on QCA evaluation

SECONDARY OUTCOMES:
Incidence of major adverse cardiac events (MACE) | 1 year, 2 years, 3 years
  Defined as a composite endpoint of all-cause death, new myocardial infarction, and unplanned revascularization
Incidence of all-cause death | 1 year, 2 years, 3 years
  Including cardiac or non-cardiac death
Incidence of new myocardial infarction | 1 year, 2 years, 3 years
Incidence of unplanned revascularization | 1 year, 2 years, 3 years
  Including infarction-related/non-infarction-related vessel revascularization
Incidence of stent thrombosis | 1 year, 2 years, 3 years
  Including probable and definite stent thrombosis
μQFR | 1 year
  Angiography-derived FFR
RWSmax, % | 1 year
  Angiography-derived radial wall strain
Diameter stenosis by QCA, % | 1 year
  Measured by QCA
Minimal fibrous cap thickness (FCTmin), mm | 1 year
  Measured by OCT
Lipid arc, ° | 1 year
  Measured by OCT
Plaque burden, % | 1 year
  Measured by OCT
Index of plaque attenuation (IPA) | 1 year
  Measured by OCT
Virtual flow ratio (VFR) | 1 year
  Measured by OCT

CONTACTS AND LOCATIONS:
Overall Officials: Lei Song, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Lei Song, Beijing, China

REFERENCES:
- [Derived] Jiang Y, Sun Z, Yu B, Liu W, Gao H, Li J, Jin Z, Yu H, Zheng B, Guan C, Zhang H, Zhang Y, Gao L, Cui C, Song Y, Xu J, Dou K, Yang W, Qian J, Wu Y, Song L. Natural history of coronary atherosclerosis based on multimodal imaging and physiological fusion techniques: study protocol and rationale for the NASCENT study. BMJ Open. 2025 Oct 23;15(10):e105796. doi: 10.1136/bmjopen-2025-105796. PMID 41130689